CLINICAL TRIAL: NCT04163458
Title: A Randomized, Double-blind Double-dummy Trial Comparing MENOPUR Solution for Injection in a Pre-filled Pen and MENOPUR Powder and Solvent for Solution for Injection (Menotropins for Injection) in a GnRH Agonist Cycle in Women Aged 18-42 Years Undergoing an Assisted Reproductive Technology Program
Brief Title: Comparison of MENOPUR Liquid and Powder in Women Undergoing Assisted Reproductive Technology (ART)
Acronym: CLARA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000303
Record Dates: First submitted 2019-10-28; First posted 2019-11-14 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-08

CONDITIONS: Infertility
Keywords: Controlled Ovarian Stimulation; Assisted Reproductive Technology
MeSH Terms: conditions — Infertility | interventions — Injections; Solvents; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MENOPUR liquid (Experimental): MENOPUR liquid (including placebo to MENOPUR powder) initiated at a fixed dose of 225 international units (IU) for first five stimulation days. From stimulation Day 6, dosing could be adjusted as needed every second day by 75 IU per adjustment based on the participant's follicular response. The maximum dose was 450 IU/day and the minimum dose was 75 IU/day. The dosing could continue for a maximum of 20 days.
  Interventions: Drug: MENOPUR solution for injection in pre-filled pen, 1200 IU/1.92 mL; Other: Placebo (for MENOPUR powder and solvent for solution for injection)
- MENOPUR powder (Active Comparator): MENOPUR powder (including placebo to MENOPUR liquid) initiated at a fixed dose of 225 IU for first five stimulation days. From stimulation Day 6, dosing could be adjusted as needed every second day by 75 IU per adjustment based on the participant's follicular response. The maximum dose was 450 IU/day and the minimum dose was 75 IU/day. The dosing could continue for a maximum of 20 days.
  Interventions: Drug: MENOPUR powder and solvent for solution for injection, 75 IU; Other: Placebo (for MENOPUR solution for injection in pre-filled pen)

INTERVENTIONS:
Drug: MENOPUR solution for injection in pre-filled pen, 1200 IU/1.92 mL — Solution for injection in pre-filled pen, subcutaneous administration
  Other Names: Highly purified menotropin
  Arms: MENOPUR liquid
Drug: MENOPUR powder and solvent for solution for injection, 75 IU — Solution for injection in vials (powder and diluent), subcutaneous administration
  Other Names: Highly purified menotropin
  Arms: MENOPUR powder
Other: Placebo (for MENOPUR solution for injection in pre-filled pen) — Solution for injection in pre-filled pen, subcutaneous administration
  Arms: MENOPUR powder
Other: Placebo (for MENOPUR powder and solvent for solution for injection) — Solution for injection in vials (powder and diluent); subcutaneous administration
  Arms: MENOPUR liquid

SUMMARY:
Development of multiple follicles and pregnancy in ovulatory women undergoing controlled ovarian stimulation as part of an assisted reproductive technology (ART) cycle.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consents, prior to any trial-related procedure.
* Females between the ages of 18 and 42 years. The participants must be at least 18 years (including the 18th birthday) when they sign the informed consent and no more than 42 years (up to the day before the 43rd birthday) at the time of randomization who desire pregnancy.
* Body mass index (BMI) between 17.5 and 38.0 kg/m^2 (both inclusive) at screening.
* Regular menstrual cycles of 24 to 35 days, presumed to be ovulatory.
* Documented history of infertility for at least 12 months before randomization for women ≤35 years or for at least 6 months for women ≥36 years. Women with documented bilateral tubal occlusion or male factor infertility requiring the use of donor sperm established as a cause of infertility are eligible at diagnosis.
* Early follicular phase (cycle day 2-4) serum FSH level between 1 and 12 IU/L (results obtained within 3 months prior to randomization).
* Male partner with semen analysis that is at least adequate for intracytoplasmic sperm injection (ICSI) at screening or within 6 months prior to the screening date. Partners with severe male factors requiring invasive or surgical sperm retrieval may not be used. Use of donor sperm is allowed.
* At least 1 cycle with no fertility medication immediately prior to screening.
* Hysterosalpingography, hysteroscopy, or saline hysterosonogram documenting uterine anatomy appropriate for ART at screening or within 12 months prior to screening.
* Transvaginal ultrasound documenting presence and adequate visualization of both ovaries, without evidence of clinically significant abnormality (e.g., endometrioma ≥3 cm, no dermoid cysts) and normal adnexa (e.g., no hydrosalpinx) at screening. Both ovaries must be accessible for oocyte retrieval.

Exclusion Criteria:

* More than two previous controlled ovarian stimulation cycles for in vitro fertilization (IVF)/ICSI
* Known stage III-IV endometriosis (American Society for Reproductive Medicine, 2012).
* Oocyte donor or embryo recipient; gestational or surrogate carrier.
* Known history of recurrent miscarriage (defined as three consecutive losses after ultrasound confirmation of pregnancy [excluding ectopic pregnancy] and before week 24 of pregnancy).
* Participant's male partner, with obvious leukospermia (>2 million white blood cells/mL) or signs of infection in semen sample within 6 months of the participant's screening. If either of these conditions exists, the male should be treated with antibiotics and retested prior to the participant's randomization.
* Active arterial or venous thromboembolism or severe thrombophlebitis, or a history of these events.
* Any known endocrine (total testosterone, prolactin and TSH) or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney) with the exception of controlled thyroid function disease.
* Known tumors of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus which would contraindicate the use of gonadotrophins.
* Any abnormal finding of clinical chemistry, hematology and vital signs at screening, which is judged clinically significant by the investigator.
* Pregnancy (negative urine pregnancy test must be documented at screening and prior to the first investigational medicinal product [IMP] administration), or contraindication to pregnancy.
* Hypersensitivity to any active ingredient or excipients in the medicinal products used in this trial.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 405 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (20):
- United States (20):
  - Fertility Treatment Center, Tempe, Arizona
  - Fertility Specialists Medical Group - San Diego Center for Reproductive Surgery, San Diego, California
  - Center for Advanced Reproductive Services PC, Farmington, Connecticut
  - Yale Fertility Center, New Haven, Connecticut
  - Fertility and IVF Center of Miami, Miami, Florida
  - Center for Reproductive Medicine, Winter Park, Florida
  - Idaho Center for Reproductive Medicine, Boise, Idaho
  - Fertility Centers of Illinois, Chicago, Illinois
  - InVia Fertility Specialists, SC, Hoffman Estates, Illinois
  - Fertility Answers, LLC, Baton Rouge, Louisiana
  - SIRM Fertility Center, Las Vegas, Nevada
  - Reproductive Endocrinology Associates of Charlotte, Charlotte, North Carolina
  - Carolina Conceptions, Raleigh, North Carolina
  - Institute for Reproductive Health, Cincinnati, Ohio
  - OU Physicians Reproductive Medicine, Oklahoma City, Oklahoma
  - Abington Reproductive Medicine, Abington, Pennsylvania
  - Fertility Associates of Memphis, PLLC, Memphis, Tennessee
  - Center for Assisted Reproduction, Bedford, Texas
  - Houston Fertility Institute, Houston, Texas
  - Center of Reproductive Medicine, Webster, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed in 19 investigational sites in US between Oct 2019 and Jul 2021.
Pre-assignment Details: In total, 691 participants were screened. Of these, 97 participants were rescreened after the trial hold was lifted, leading to a total of 788 screening events. Of these, 383 were screening event failures while 405 screening events resulted in randomization. 401 participants were exposed to IMP: 202 participants exposed to MENOPUR liquid and 199 participants were exposed to MENOPUR powder.
Period: Overall Study
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Started | 204 | 201
mITT | 202 | 199
Completed | 180 | 171
Not Completed | 24 | 30
Not completed — Protocol Deviation | 7 | 13
Not completed — Adverse Event | 5 | 8
Not completed — Due to COVID-19 pandemic | 4 | 2
Not completed — Participant withdrew consent | 2 | 3
Not completed — Randomization failure | 2 | 2
Not completed — Other | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MENOPUR Liquid | MENOPUR Powder | Total
Number analyzed (Participants) | 202 | 199 | 401
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.9 (3.9) | 34.0 (4.3) | 34.0 (4.1)
Age, Customized [Count of Participants; unit: Participants]
  Age: <35 years | 111 | 107 | 218
  Age: >=35 years | 91 | 92 | 183
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 199 | 401
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 26 | 60
  Not Hispanic or Latino | 168 | 173 | 341
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 17 | 16 | 33
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 23 | 19 | 42
  White | 158 | 160 | 318
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 202 | 199 | 401
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (4.6) | 25.9 (4.7) | 26.0 (4.7)
Primary Infertility [Count of Participants; unit: Participants]
  Yes | 102 | 102 | 204
  No | 100 | 97 | 197
Duration of infertility [Mean (Standard Deviation); unit: Months] | 46.1 (36.8) | 44.5 (31.4) | 45.3 (34.2)
Primary reason for infertility [Count of Participants; unit: Participants]
  Unexplained infertility | 91 | 79 | 170
  Tubal infertility | 40 | 39 | 79
  Mild male factor | 17 | 27 | 44
  Moderate male factor | 24 | 24 | 48
  Severe male factor | 21 | 25 | 46
  Endometriosis stage I/II | 9 | 4 | 13
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Fertilized (2 Pronuclei [2PN]) Oocytes
Description: Fertilized oocytes with 2PN were regarded as correctly fertilized.
Time Frame: On Day 1 after oocyte retrieval (up to 23 days after start of stimulation)
Measure: Mean (Standard Deviation); unit: Fertilized oocytes
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Fertilized oocytes | 8.3 (5.5) | 6.7 (4.2)

2. Secondary Outcome: Positive Beta Human Chorionic Gonadotropin (βhCG) Rate
Description: A blood serum βhCG test was obtained 10-14 days after blastocyst transfer. If the test was positive according to the local laboratory's reference ranges, this confirmed a positive βhCG.
Time Frame: 10-14 days after blastocyst transfer (up to approximately 6 weeks after start of stimulation)
Measure: Count of Participants; unit: Participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Participants | 113 | 110

3. Secondary Outcome: Clinical Pregnancy Rate
Description: Clinical pregnancy was based on detection of at least 1 intrauterine gestational sac with fetal heart beat on transvaginal ultrasound.
Time Frame: 5-6 weeks after blastocyst transfer (up to approximately 10 weeks after start of stimulation)
Measure: Count of Participants; unit: Participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Participants | 94 | 88

4. Secondary Outcome: Ongoing Pregnancy Rate
Description: Ongoing pregnancy was based on detection of at least 1 intrauterine viable fetus by transvaginal or abdominal ultrasound
Time Frame: 8-9 weeks after blastocyst transfer (up to approximately 13 weeks after start of stimulation)
Measure: Count of Participants; unit: Participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Participants | 91 | 85

5. Secondary Outcome: Early Pregnancy Loss
Description: Number of participants with early pregnancy loss defined as a positive βhCG tests but no ongoing pregnancy.
Time Frame: 8-9 weeks after blastocyst transfer (up to approximately 13 weeks after start of stimulation)
Population: Only participants who had a positive βhCG test were eligible.
Measure: Count of Participants; unit: Participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 113 | 110
Participants | 22 | 25

6. Secondary Outcome: Follicular Development on Stimulation Day 6
Description: The total number of follicles and the number of follicles per size category were reported.
Time Frame: At stimulation Day 6
Measure: Mean (Standard Deviation); unit: Follicles
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Follicles
  Total number of follicles | 17.0 (9.4) | 16.5 (8.3)
  Follicles >= 12 mm | 1.8 (2.3) | 1.5 (2.0)
  Follicles >= 15 mm | 0.2 (0.6) | 0.2 (0.6)
  Follicles >= 17 mm | 0.0 (0.2) | 0.0 (0.1)

7. Secondary Outcome: Follicular Development on Last Day of Stimulation
Description: The total number of follicles and the number of follicles per size category were reported.
Time Frame: At last day of stimulation (up to 20 stimulation days)
Measure: Mean (Standard Deviation); unit: Follicles
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Follicles
  Total number of follicles | 19.9 (9.8) | 19.2 (10.1)
  Follicles >= 12 mm | 13.1 (5.2) | 12.0 (5.1)
  Follicles >= 15 mm | 8.5 (3.1) | 8.1 (3.2)
  Follicles >= 17 mm | 5.4 (2.3) | 5.2 (2.2)

8. Secondary Outcome: Serum Follicle-stimulating Hormone (FSH) Concentration
Description: The concentration of serum FSH was measured. The median and IQR of FSH levels on stimulation day 6, End of stimulation and Oocyte Retrieval visit are presented.
Time Frame: At Day 6, last day of stimulation (up to 20 stimulation days) and at oocyte retrieval (up to 22 days after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 201 | 198
IU/L
  Stimulation Day 6: number analyzed (Participants) | 200 | 198
  Stimulation Day 6 | 16.7 [14.1 to 20.2] | 14.9 [12.8 to 17.2]
  End of stimulation: number analyzed (Participants) | 201 | 192
  End of stimulation | 17.6 [13.9 to 22.5] | 16.5 [13.8 to 20.5]
  Oocyte retrieval: number analyzed (Participants) | 189 | 184
  Oocyte retrieval | 8.8 [7.1 to 12.3] | 8.4 [6.7 to 10.5]

9. Secondary Outcome: Serum Anti-Müllerian Hormone (AMH) Concentration
Description: The concentration of serum AMH was measured. The median and IQR of AMH levels on End of stimulation and End of Trial are presented.
Time Frame: At the last day of stimulation (up to 20 stimulation days) and at end-of-trial (up to approximately 6 months from the start of screening)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 201 | 192
pmol/L
  End of stimulation | 7.6 [5.4 to 12.3] | 8.7 [5.6 to 12.9]
  End of trial: number analyzed (Participants) | 195 | 190
  End of trial | 16.5 [10.1 to 24.0] | 15.5 [11.1 to 22.1]

10. Secondary Outcome: Human Chorionic Gonadotropin (hCG) Concentration
Description: The concentration of hCG was measured. The median and IQR of hCG levels on stimulation day 6 and End of stimulation are presented.
Time Frame: At Day 6 and last day of stimulation (up to 20 stimulation days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 201 | 198
IU/L
  Stimulation Day 6: number analyzed (Participants) | 200 | 198
  Stimulation Day 6 | 2.5 [2.0 to 3.1] | 2.4 [1.9 to 2.9]
  End of stimulation: number analyzed (Participants) | 201 | 192
  End of stimulation | 2.7 [1.9 to 3.5] | 2.7 [2.1 to 3.4]

11. Secondary Outcome: Luteinizing Hormone (LH) Concentration
Description: The concentration of LH was measured. The median and IQR of LH levels on stimulation day 6 and End of stimulation are presented.
Time Frame: At Day 6 and last day of stimulation (up to 20 stimulation days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 201 | 198
IU/L
  Stimulation Day 6: number analyzed (Participants) | 200 | 198
  Stimulation Day 6 | 1.8 [1.2 to 2.4] | 1.8 [1.2 to 2.4]
  End of stimulation: number analyzed (Participants) | 201 | 192
  End of stimulation | 3.3 [2.2 to 4.3] | 3.1 [2.2 to 4.4]

12. Secondary Outcome: Progesterone (P4) Concentration
Description: The concentration of P4 was measured. The median and IQR of P4 levels on stimulation day 6 and End of stimulation are presented.
Time Frame: At Day 6 and last day of stimulation (up to 20 stimulation days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 201 | 198
ng/mL
  Stimulation Day 6: number analyzed (Participants) | 200 | 198
  Stimulation Day 6 | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.4]
  End of stimulation: number analyzed (Participants) | 201 | 192
  End of stimulation | 0.8 [0.6 to 1.1] | 0.6 [0.4 to 1.0]

13. Secondary Outcome: Estradiol (E2) Concentration
Description: The concentration of E2 was measured. The median and IQR of E2 levels on stimulation day 6 and End of stimulation are presented.
Time Frame: At stimulation Day 6 and last day of stimulation (up to 20 stimulation days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 201 | 198
pg/mL
  Stimulation Day 6: number analyzed (Participants) | 200 | 198
  Stimulation Day 6 | 518.1 [236.7 to 834.0] | 336.4 [167.5 to 607.2]
  End of stimulation: number analyzed (Participants) | 201 | 192
  End of stimulation | 2720.0 [1994.0 to 3266.0] | 2292.0 [1694.0 to 2887.5]

14. Secondary Outcome: Number of Oocytes Retrieved
Description: The number of oocytes retrieved was recorded at the oocyte retrieval visit.
Time Frame: On day of oocyte retrieval (up to 22 days after start of stimulation)
Measure: Mean (Standard Deviation); unit: Oocytes
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Oocytes | 14.3 (8.1) | 11.4 (6.3)

15. Secondary Outcome: Number of Metaphase II (MII) Oocytes
Description: Maturity stage was assessed prior to undergoing ICSI. Maturity stage was categorized as germinal vesicle, metaphase I, metaphase II, degenerated or other.
Time Frame: On day of oocyte retrieval (up to 22 days after start of stimulation)
Population: Only participants with Oocytes retrieved were eligible.
Measure: Mean (Standard Deviation); unit: MII Oocytes
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 199 | 189
MII Oocytes | 10.6 (6.1) | 8.9 (4.8)

16. Secondary Outcome: Fertilization Rate
Description: Fertilization rate(%) is the number of 2PN oocytes divided by the number of oocytes retrieved.
Time Frame: On Day 1 after oocyte retrieval (up to 23 days after start of stimulation)
Population: Only participants with Oocytes retrieved were eligible.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 199 | 189
Percentage | 57.8 (19.9) | 60.0 (20.9)

17. Secondary Outcome: Number of Blastocysts and Number of Good-Quality Blastocysts 5 Days After Oocyte Retrieval
Description: The number of blastocysts (total and good-quality) was reported. Blastocyst quality was assessed by blastocyst expansion and hatching status, blastocyst inner cell mass grading, and trophectoderm grading. The scoring was based on the classification system by Gardner and Schoolcraft, with additional categories for inner cell mass (degenerative or no inner cell mass) and trophectoderm (degenerative or very large cells)
Time Frame: On Day 5 after oocyte retrieval (up to 27 days after start of stimulation)
Measure: Mean (Standard Deviation); unit: Blastocysts
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Blastocysts
  Number of Blastocysts on Day 5 | 4.8 (3.8) | 3.9 (3.0)
  Number of Good-quality blastocysts on Day 5 | 3.0 (3.0) | 2.6 (2.6)

18. Secondary Outcome: Total Gonadotropin Dose
Description: The gonadotropin starting dose was 225 IU for the first 5 days, followed by individual adjustments according to the participant's follicular response. Dose adjustment should be 75 IU per adjustment. Gonadotropin was to be initiated within 3 days of confirmed downregulation.
Time Frame: Up to 20 stimulation days
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
IU | 2265.6 (710.2) | 2466.7 (863.5)

19. Secondary Outcome: Number of Stimulation Days
Description: Calculated by start dates and end dates.
Time Frame: Up to 20 stimulation days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Days | 9.6 (1.7) | 9.9 (1.8)

20. Secondary Outcome: Proportion of Participants With Ovarian Hyperstimulation Syndrome (OHSS)
Description: OHSS was defined as the total of early OHSS with onset ≤9 days after triggering of final follicular maturation, and late OHSS with onset >9 days after triggering of final follicular maturation.
Time Frame: ≤9 days after triggering of final follicular maturation (early OHSS), >9 days after triggering of final follicular maturation until 21-28 days after last IMP dose or up to ongoing pregnancy 8-9 weeks after transfer in pregnant participants (late OHSS)
Measure: Number; unit: Percentage of participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Percentage of participants
  Early OHSS | 3.5 | 3.5
  Late OHSS | 4.0 | 1.5

21. Secondary Outcome: Frequency of Adverse Events (AEs)
Description: Any AE occurring after start of IMP and before the end-of-trial visit, or a pre-treatment AE or pre-existing medical condition that worsens in intensity after start of IMP and before the end-of-trial visit was considered treatment-emergent, and is presented for this endpoint.
Time Frame: From the time of signed informed consent for participation in the trial until the end-of-trial visit (up to approximately 6 months)
Measure: Number; unit: Percentage of participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Percentage of participants | 50.0 | 52.3

22. Secondary Outcome: Intensity of AEs
Description: The intensity of an AE was classified using the following 3-point scale: Mild = Awareness of signs or symptoms, but no disruption of usual activity. Moderate = Event sufficient to affect usual activity (disturbing). Severe = Inability to work or perform usual activities (unacceptable).
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Measure: Number; unit: Percentage of participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Percentage of participants
  Mild AEs | 42.1 | 40.7
  Moderate AEs | 23.8 | 20.6
  Severe AEs | 0.5 | 2.0

23. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Alanine Aminotransferase
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
IU/L | 0.4 (14.2) | -1.0 (12.4)

24. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Aspartate Aminotransferase
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
IU/L | -0.9 (8.8) | -2.1 (21.1)

25. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Blood Urea Nitrogen
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
mmol/L | -0.7 (1.2) | -0.7 (1.3)

26. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Calcium
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
mmol/L | -0.03 (0.10) | -0.03 (0.08)

27. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Chloride
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
mmol/L | 0.4 (2.3) | 0.3 (2.2)

28. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
umol/L | -5.498 (10.896) | -5.032 (8.849)

29. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Gamma Glutamyl Transferase
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
IU/L | -0.6 (5.6) | -1.6 (8.9)

30. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Glucose
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
mmol/L | 0.0 (0.8) | -0.1 (0.9)

31. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Potassium
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
mmol/L | -0.04 (0.38) | -0.05 (0.40)

32. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Sodium
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 196 | 185
mmol/L | -1.0 (3.0) | -0.8 (3.1)

33. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Egfr African American
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 23 | 19
mL/min/1.73m2 | 7.7 (14.9) | 2.4 (13.7)

34. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Parameters Compared to Baseline: Egfr Non-afr. American
Description: Blood samples were collected for the analysis of clinical chemistry parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 173 | 166
mL/min/1.73m2 | 6.3 (13.1) | 5.9 (11.6)

35. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Erythrocytes
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
10^12 cells/L | -0.169 (0.293) | -0.199 (0.256)

36. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Leukocytes
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
10^9 cells/L | 1.17 (2.25) | 1.11 (2.09)

37. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Hemoglobin
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
g/L | -4.40 (9.87) | -5.76 (8.02)

38. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Hematocrit
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: RATIO
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
RATIO | -0.02 (0.03) | -0.02 (0.03)

39. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Platelets
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 182
10^9 cells/L | 22.6 (38.6) | 23.7 (43.2)

40. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Basophils
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
cells/uL | 1.7 (54.0) | -0.1 (60.6)

41. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Basophils/Leukocytes
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Basophils/leukocytes in Percentage
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
Basophils/leukocytes in Percentage | -0.1 (0.8) | -0.2 (1.0)

42. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Eosinophils
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
cells/uL | -10.6 (100.5) | 4.2 (68.6)

43. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Eosinophils/Leukocytes
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Eosinophils/leukocytes in percentage
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
Eosinophils/leukocytes in percentage | -0.4 (1.6) | -0.1 (1.2)

44. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Lymphocytes
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
cells/uL | -53.2 (414.9) | -4.0 (442.5)

45. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Lymphocytes/Leukocytes
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lymphocytes/leukocytes in percentage
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
Lymphocytes/leukocytes in percentage | -4.5 (9.6) | -3.4 (9.5)

46. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Monocytes
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
cells/uL | 21.5 (161.8) | 36.7 (148.9)

47. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Monocytes/Leukocytes
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Monocytes/leukocytes in percentage
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
Monocytes/leukocytes in percentage | -0.8 (1.7) | -0.5 (1.6)

48. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Neutrophils
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
cells/uL | 1206.4 (2096.6) | 1069.0 (1966.0)

49. Secondary Outcome: Changes in Circulating Levels of Haematology Parameters Compared to Baseline: Neutrophils/Leukocytes
Description: Blood samples were collected for the analysis of haematology parameters.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Neutrophils/leukocytes in percentage
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 197 | 183
Neutrophils/leukocytes in percentage | 5.7 (11.2) | 4.2 (10.6)

50. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Changes of Clinical Parameters and Haematology Parameters
Description: The table represents the percentage of participants in each group with normal baseline values and markedly abnormal end-of-stimulation or end-of-trial visit values.
  It is only parameters with markedly abnormal values at end of stimulation or end of trial visit which are represented. Parameters with normal baseline values and normal end of stimulation and end of trial values are not represented.
Time Frame: From the start of screening until the end-of-trial (up to approximately 6 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure. Participants who were evaluable had normal baseline values and markedly abnormal end-of-stimulation or end-of-trial visit values.
Measure: Count of Participants; unit: Participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 198 | 189
Participants
  Calcium (mmol/L) (End of stimulation): number analyzed (Participants) | 194 | 183
  Calcium (mmol/L) (End of stimulation) | 1 | 0
  Glucose (mmol/L) (End of stimulation) | 1 | 0
  Erythrocytes (10^12 cells/L) (End of stimulation): number analyzed (Participants) | 185 | 183
  Erythrocytes (10^12 cells/L) (End of stimulation) | 2 | 0
  Leukocytes (10^9 cells/L) (End of stimulation): number analyzed (Participants) | 189 | 175
  Leukocytes (10^9 cells/L) (End of stimulation) | 2 | 0
  Hemoglobin (g/L) (End of stimulation): number analyzed (Participants) | 190 | 184
  Hemoglobin (g/L) (End of stimulation) | 2 | 0
  Hematocrit (RATIO) (End of stimulation): number analyzed (Participants) | 179 | 178
  Hematocrit (RATIO) (End of stimulation) | 2 | 0
  Platelets (10^9 cells/L) (End of stimulation): number analyzed (Participants) | 191 | 181
  Platelets (10^9 cells/L) (End of stimulation) | 1 | 0
  Basophils/leukocytes ratio (%) (End of stimulation): number analyzed (Participants) | 182 | 172
  Basophils/leukocytes ratio (%) (End of stimulation) | 1 | 0
  Lymphocytes/leukocytes ratio (%) (End of stimulation): number analyzed (Participants) | 189 | 185
  Lymphocytes/leukocytes ratio (%) (End of stimulation) | 2 | 0
  Alanine Aminotransferase (IU/L) (End of trial): number analyzed (Participants) | 185 | 175
  Alanine Aminotransferase (IU/L) (End of trial) | 1 | 0
  Leukocytes (10^9 cells/L) (End of trial): number analyzed (Participants) | 190 | 169
  Leukocytes (10^9 cells/L) (End of trial) | 1 | 1

51. Secondary Outcome: Frequency of Injection Site Reactions (Redness, Pain, Itching, Swelling and Bruising) Assessed by the Participant During the Stimulation Period
Description: Assessed by the participant during the stimulation period. Participants assessed the injection site reactions (redness, pain, itching, swelling and bruising) three times daily: immediately after the injection, 30 minutes after the injection and 24 hours after the injection.
  Total Number of events include all categories None, Mild, Moderate and Severe. Percentage of events with injection site reactions as a sum of the categories Mild, Moderate and Severe is presented.
Time Frame: Up to 20 stimulation days
Measure: Number; unit: Percentage of events
Units Other Than Participants: Total number of events
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Number analyzed (Total number of events) | 29185 | 29425
Percentage of events | 6.3 | 14.5

52. Secondary Outcome: Intensity of Injection Site Reactions (Redness, Pain, Itching, Swelling and Bruising) Assessed by the Participant During the Stimulation Period
Description: Assessed by the participant during the stimulation period as mild, moderate or severe.
  Participants assessed the injection site reactions (redness, pain, itching, swelling and bruising) three times daily: immediately after the injection, 30 minutes after the injection and 24 hours after the injection.
Time Frame: Up to 20 stimulation days
Measure: Number; unit: Percentage of events
Units Other Than Participants: Total number of events
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Number analyzed (Total number of events) | 29185 | 29425
Percentage of events
  Mild injection site reaction | 6.1 | 12.9
  Moderate injection site reaction | 0.2 | 1.4
  Severe injection site reaction | 0.0069 | 0.2

53. Secondary Outcome: Proportion of Participants With Treatment-induced Anti-MENOPUR Antibodies. Overall as Well as With Neutralizing Capacity
Description: Measured by presence of anti-MENOPUR antibodies.
  95% Clopper-Pearson confidence interval has been reported in this endpoint.
Time Frame: Up to 28 days after end of the stimulation period (simulation period up to 20 days)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Percentage of participants
  Treatment-induced anti-MENOPUR antibodies (overall) | 1.5 [0.3 to 4.3] | 1.5 [0.3 to 4.3]
  Treatment-induced anti-MENOPUR antibodies with neutralizing capacity | 0 [0 to 1.81] | 0 [0 to 1.84]

54. Secondary Outcome: Number of Participants With Potential Technical Malfunctions of the Administration Pen
Description: Number of participants With Potential Technical malfunctions of the Administration Pen were recorded.
Time Frame: Up to 20 stimulation days
Measure: Count of Participants; unit: Participants
Arm/Group | MENOPUR Liquid | MENOPUR Powder
Number analyzed (Participants) | 202 | 199
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of signed informed consent for participation in the trial until the end-of-trial visit (up to approximately 6 months).
Arm/Group | MENOPUR Liquid | MENOPUR Powder
All-Cause Mortality (participants affected / at risk) | 0/202 | 0/199
Serious Adverse Events (participants affected / at risk) | 4/202 | 2/199
Other Adverse Events (participants affected / at risk) | 101/202 | 104/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MENOPUR Liquid (N=202) | MENOPUR Powder (N=199)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 4 (4) | 2 (2)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MENOPUR Liquid (N=202) | MENOPUR Powder (N=199)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 7 (7)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 39 (40) | 38 (38)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 6 (6) | 12 (13)
Migraine (Nervous system disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 18 (22) | 22 (26)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 11 (11)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 13 (13)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 5 (5)
Subchorionic haemorrhage (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
Subchorionic haematoma (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 3 (3)
Pelvic discomfort (Reproductive system and breast disorders) | 17 (19) | 10 (13)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 15 (15) | 10 (10)
Pelvic pain (Reproductive system and breast disorders) | 14 (15) | 8 (9)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT04163458/Prot_002.pdf
  • Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT04163458/SAP_001.pdf